CLINICAL TRIAL: NCT05437471
Title: Effects of Co-treatment With Aromatase Inhibitor or Progestin on Endometrial abv3-integrin Expressions in Women With Recurrent Implantation Failure
Brief Title: Effects of Co-treatment on Endometrial abv3-integrin Expressions in Women With Recurrent Implantation Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Thines Ramalingam, Doctor, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GGPM-2019-034
Record Dates: First submitted 2022-03-29; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Miscarriage, Recurrent
MeSH Terms: conditions — Abortion, Habitual | interventions — Dydrogesterone; Letrozole

STUDY DESIGN:
Intervention Model Description: All recruited women will be allocated in three groups, and endometrial tissue sampling will be obtained prior to medical intervention assigned during luteal phase depending on their menstrual cycle. All these women will be divided randomly in three groups A, B & C equally by using the auto-randomized program in SPSS version 21.0.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (GnRH analogue with Aromatase Inhibitor (Active Comparator): This group of candidates will be administered a single dose of 11.25mg GNRH analoge (Lucrin) followed by Letroloze 10mg OD for 3 months
  Interventions: Drug: GNRH Analoge, Duphaston, Letrozole
- Group B (GnRH analogue with Progesterone (Active Comparator): This group of candidates will be administered a single dose of 11.25mg GNRH analoge (Lucrin) followed Duphaston 10mg BD by for 3 months
  Interventions: Drug: GNRH Analoge, Duphaston, Letrozole
- Group C (GnRH analogue alone) (Placebo Comparator): This is a control group. The candidates will be administered a single dose of 11.25mg GNRH analoge (Lucrin) only.
  Interventions: Drug: GNRH Analoge, Duphaston, Letrozole

INTERVENTIONS:
Drug: GNRH Analoge, Duphaston, Letrozole — GNRH Analoge, Duphaston, Letrozole

SUMMARY:
To compare the abv3-integrin expression in endometrium tissue among RIF women between the GnRH analogue with Aromatase Inhibitor (Group A) , GnRH analogue with progesterone (Group B) and GnRH analogue alone as control group (Group C)

DETAILED DESCRIPTION:
i. To determine the abv3-integrin expression isolated from endometrium tissue from women with RIF prior to medical therapy.

ii. To determine the abv3-integrin expression isolated from endometrium tissue from Group A, Group B and Group C following the medical therapy.

iii. To compare the abv3-integrin expression from endometrium tissue obtained from Group A, B and C following the medical therapy.

iv. To compare the implantation rates among Group A, B and C following the medical therapy.

v. To compare the ongoing pregnancy among Group A, B and C following the medical therapy

ELIGIBILITY:
Inclusion Criteria:

* Women of 18 to 40 years of age
* No significant pre-existing major medical.
* Diagnosed as recurrent implantation failure - at least two or more failure of achieving pregnancy following embryo transfer (ET) despite the optimum endometrial thickness and good quality of embryo (unexplained).
* Regular menstrual cycle atleast 3 months prior to treatment
* Not taking any hormonal treatment for atlest 3months prior to recruitment
* Agreed to participate

Exclusion Criteria:

* Concurrent significant pre-existing major medical conditions such as uncontrolled diabetes, active systemic lupus erythematosus (SLE) or Anti Phospholipid Syndrome (APS) that will interfere with implantation.
* Poor quality of embryo
* Suboptimal endometrial thickness(<8mm) during the embryo transfer (ET).
* On hormonal therapy prior to recruitment.
* Not agreed to participate

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
endometrial abv3-integrin expression expressions | 12 months
  pre and post treatment endometrial abv3-integrin expressions

CONTACTS AND LOCATIONS:
Locations (1):
- UniversitiKMMC, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided